CLINICAL TRIAL: NCT02151734
Title: Safety and Efficacy of KALOMIN™ Tab. in Patients With Acute Bronchitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KUP-KLM_301
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Acute Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- KALOMIN™ Tab. (Experimental): KALOMIN™ Tab./Placebo to Umckamin syrup
  Interventions: Drug: KALOMIN™ Tab.
- Umckamin syrup (Active Comparator): Umckamin syrup/Placebo to KALOMIN™ Tab.
  Interventions: Drug: Umckamin syrup

INTERVENTIONS:
Drug: KALOMIN™ Tab.
  Arms: KALOMIN™ Tab.
Drug: Umckamin syrup
  Arms: Umckamin syrup

SUMMARY:
This is a multi-center, double-dummy, double-blind, randomized, active-controlled, parallel group phase 3 clinical trial to evaluate the efficacy and safety of KALOMIN™ Tab. in patients with acute bronchitis.

The aim of this clinical trial is to demonstrate that KALOMIN™ Tab. is clinically non-inferior to Umckamin syrup, as assessed by BSS(Bronchitis Severity Score), in the treatment of acute bronchitis after 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 12-75 years old
* A total score of BSS ≥ 5
* The duration of symptoms had to be less than 14 days and no chronic pulmonary disease
* Patients who voluntarily sign a written informed consent to participate in the trial

Exclusion Criteria:

* Indication for antibiotic treatment(e.g. severe respiratory infection)
* Allergic bronchial asthma
* Tendency to bleed
* Severe heart, renal, or liver diseases or decline of immune function
* Chronic obstructive pulmonary disease
* Known or supposed hypersensitivity to investigational medication
* Treatment with antibiotics during the past 4 weeks prior to inclusion in the trial
* Women during pregnancy or lactation period
* Clinically significant abnormal values in the screening test(more than twice the upper limit of normal range for ALT, AST, BUN, and Serum Creatinine)
* Participation in any other trial within 30 days prior to inclusion in the trial
* Unsuitable patients for enrollment in the opinion of the investigator

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Total score of BSS(Bronchitis Severity Score) | 7days

SECONDARY OUTCOMES:
Individual symptom score of BSS | 7days
reaction rate of treatment | 7days
IMOS(Integrative Medicine Outcome Scale) | 7days
IMPSS(Integrative Medicine Patient Satisfaction Scale) | 7days
Adverse events, clinical laboratory examination, physical examination, etc. | 7 days